CLINICAL TRIAL: NCT02330770
Title: Dual Trigger Versus Gonadotropin Releasing Hormone Agonist Trigger Combined With Luteal Human Chorionic Gonadotropin Administration
Brief Title: Dual Trigger Versus GnRHa Trigger Combined With Luteal HCG Administration
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Sayed Abdelhafez, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MSA5
Record Dates: First submitted 2015-01-01; First posted 2015-01-05 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Infertility
Keywords: GnRHa trigger; Luteal phase support; OHSS
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate; Chorionic Gonadotropin; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dual trigger group (Active Comparator): Trigger with concomitant GnRHa and HCG (single low-dose) administration
  Interventions: Drug: GnRHa and HCG
- Single low-dose HCG group (Active Comparator): Trigger with GnRHa then HCG (single low-dose) administration in luteal phase
  Interventions: Drug: GnRHa then HCG (single low-dose)
- Multiple low-doses HCG group (Active Comparator): Trigger with GnRHa then HCG (multiple low-doses) administration in luteal phase
  Interventions: Drug: GnRHa then HCG (multiple low-doses)

INTERVENTIONS:
Drug: GnRHa and HCG — Final oocyte maturation will be triggered by dual administration of 0.2 mg of GnRHa preparation (Triptorelin) SC and 1500 IU of HCG preparation IM
  Other Names: Decapeptyl and Pregnyl
  Arms: Dual trigger group
Drug: GnRHa then HCG (single low-dose) — Final oocyte maturation will be triggered by administration of 0.2 mg Triptorelin SC then a single IM bolus of 1500 IU HCG will be administered 35-37 hours after GnRHa trigger (1 hour after oocyte retrieval)
  Other Names: Decapeptyl then Pregnyl
  Arms: Single low-dose HCG group
Drug: GnRHa then HCG (multiple low-doses) — Final oocyte maturation will be triggered by administration of 0.2 mg Triptorelin SC then 3 IM boluses of 500 IU HCG will be administered day 1, day 4 and day 7 after oocyte retrieval
  Other Names: Decapeptyl then Pregnyl
  Arms: Multiple low-doses HCG group

SUMMARY:
Comparing the reproductive outcomes of intracytoplasmic sperm injection (ICSI) cycles in women at risk of ovarian hyperstimulation syndrome (OHSS) subjected to gonadotropin releasing hormone (GnRH) antagonist protocol followed by trigger with concomitant GnRH agonist (GnRHa) and low-dose human chorionic gonadotropin (HCG) administration (dual trigger), GnRHa trigger with single luteal low-dose HCG or GnRHa trigger with multiple luteal low-doses HCG

DETAILED DESCRIPTION:
The GnRH antagonist fixed protocol will be used for controlled ovarian hyperstimulation (COH). Transvaginal sonography (TVS) scan will be performed regularly for monitoring of the follicular growth (folliculometry). When there will be at least 3 leading follicles > 18 mm in diameter, women will be randomized into 3 groups; group A (dual trigger group), group B (single low-dose HCG group) and group C (multiple low-doses HCG group). In group A, final oocyte maturation will be triggered by dual administration of 0.2 mg of GnRHa preparation (Triptorelin) SC and 1500 IU of HCG preparation IM. In group B, final oocyte maturation will be triggered by administration of 0.2 mg Triptorelin SC then a single IM bolus of 1500 IU HCG will by administered 35-37 hours after GnRHa trigger (1 hour after oocyte retrieval). In group C, final oocyte maturation will be triggered by administration of 0.2 mg Triptorelin SC then 3 IM boluses of 500 IU HCG will be administered day 1, day 4 and day 7 after oocyte retrieval. In all women, oocyte retrieval will be performed 34-36 hours after trigger and endometrial preparation for embryo transfer (ET) will be started on the day of oocyte retrieval by giving 400 mg vaginal natural progesterone supplement once daily plus 4 mg oral estradiol valerate once daily.

ELIGIBILITY:
Inclusion Criteria:

* Women subjected to ICSI through controlled ovarian hyperstimulation (COH) with pituitary downregulation by GnRH antagonist.
* Presence of risk for development of OHSS: 1) previous moderate or severe OHSS; 2) PCOS or polycystic ovary on ultrasound scan; 3) antral follicle count (AFC) > 14 in both ovaries; 4) basal serum AMH level > 3.36 ng/ml; 5) > 14 follicles with diameter of ≥ 11 mm on the day of triggering of oocyte maturation; 6) E2 level > 3000 pg/ml on the day of triggering of oocyte maturation.

Exclusion Criteria:

* Age < 20 years or > 35 years.
* BMI < 19 kg/m2 or > 35 kg/m2.
* Moderate or severe endometriosis.
* Hydrosalpinx.
* Uterine abnormalities or myoma.
* Previous uterine surgery.
* Use of alternative techniques to minimize the risk of OHSS.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 225 (Estimated)
Dates: Start 2016-06-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6 weeks after embryo transfer
  Number of clinical pregnancies (defined as presence of at least one intrauterine gestational sac with fetal pole and cardiac activity on TVS scan at 4-6 weeks after the ET) divided by the number of ET procedures

SECONDARY OUTCOMES:
Oocyte maturation rate | On day of oocyte retrieval
  Number of mature oocytes divided by the number of retrieved oocytes
Incidence of early OHSS | Within 9 days of final triggering of oocyte maturation
  Incidence of OHSS within 9 days of final triggering of oocyte maturation
Implantation rate | 6 weeks after embryo transfer
  Number of gestational sacs on TVS scan at 4-6 weeks after ET divided by the number of transferred embryos
Miscarriage rate | 12 weeks gestational age
  Number of first trimester miscarriages (before 12 weeks gestational age) divided by the number of clinical pregnancies

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Abdelhafez, Dr, Principal Investigator — Mansoura University; Waleed El-refaie, Dr, Study Director — Port Said University
Locations (2):
- Egypt (2):
  - Fertility Care Unit (FCU) in Mansoura University Hospital, Al Mansurah, Dakahlia Governorate
  - Private fertility care centers, Al Mansurah, Dakahlia Governorate

IPD SHARING:
Plan to Share IPD: No